CLINICAL TRIAL: NCT05830006
Title: Indications and Evaluation of Microfat Grafting in Cleft Lip Nasal Deformities
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Susanna Nabil Habib, Principal Investigator Resident doctor at plastic and reconstructive surgery department at elmabbara health insurance hospital, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Microfat grafting in nose
Record Dates: First submitted 2022-04-22; First posted 2023-04-26 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Cleft Lip and Nose
Keywords: microfat grafting
MeSH Terms: conditions — Cleft Lip

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- main group (Experimental)
  Interventions: Procedure: Microfat grafting

INTERVENTIONS:
Procedure: Microfat grafting — Microfat grafting in cleft lip nasal deformities

SUMMARY:
Aim of the work:

The study will be conducted to investigate the efficacy of microfat graftinig in cleft lip nasal deformities especially in young patients and those adults who don't need major correction after rhinoplasty.

DETAILED DESCRIPTION:
Microfat grafting was used for the first time in 1880, in reconstructive surgery to correct facial deformities, to reconstruct defects post oncological surgery, to treat complex wounds, and to manage scars. Therefore its usage is increasing widely and particularly in maxillofacial and plastic surgeries.

As lipofilling is a potential filler of reference for rhinoplasty and it can be performed on the dorsum, radix, glabella, pre-maxilla, and nasal pyramid. The investigators are suggesting it's use in cleft lip nasal deformities in some special situations.

Imperfections post rhinoplasty are common and there is an increased risk of patient dissatisfaction in revision surgeries. This may be due to a change in the nasal anatomy, the development of scar tissue, the loss of cartilaginous support, the altered blood supply, and the compromised soft tissue envelope. Here comes the role of fat grafting which is a relatively simple and safe procedure to camouflage nose imperfections in filling the subcutaneous tissue, and in improving the skin quality post rhinoplasty.

Microfat grafting appears to be effective for correcting minor irregularities of nasal skin and may be appropriate for patients who cannot undergo revision rhinoplasty. It is also an effective salvage procedure for severely damaged skin of the nose. Injection of cryopreserved fat over several sessions is well accepted by patients because cryopreservation of excess harvested fat grafts for subsequent use makes repeated fat graft harvesting unnecessary. Microfat grafting is not a replacement for, but may be a complement to, modern rhinoplasty techniques.

ELIGIBILITY:
Inclusion Criteria:

1. Gender : Both sex will be included in the study.
2. Postcleft lip nose deformities.

Exclusion Criteria:

1. Refusing enrollment into the study.
2. Refusing the surgery.
3. Contraindication to anaesthesia.

Ages: 5 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Anthropometric measurement for the nose in relation to face | 6 months
  Results would be depending on objective and subjective measures :
  *Objective assessment by taking photos by anthropometric measurement for the nose in relation to face.

SECONDARY OUTCOMES:
patient and thier parents satisfaction | 6 months
  *Subjective assessment by evaluate patients & their parents satisfaction from the result
  From zero to 4 as :
  Zero = not satisfied
  1. = fair satisfaction
  2. = good
  3. = very good
  4. = fully satisfied Higher scores means better

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Ali, lecturer, Study Chair — Assiut University

REFERENCES:
- [Background] Simonacci F, Bertozzi N, Grieco MP, Grignaffini E, Raposio E. Procedure, applications, and outcomes of autologous fat grafting. Ann Med Surg (Lond). 2017 Jun 27;20:49-60. doi: 10.1016/j.amsu.2017.06.059. eCollection 2017 Aug. PMID 28702187
- [Background] Benateau H, Rocha CS, Rocha Fde S, Veyssiere A. Treatment of the nasal abnormalities of Hallermann-Streiff syndrome by lipofilling. Int J Oral Maxillofac Surg. 2015 Oct;44(10):1246-9. doi: 10.1016/j.ijom.2015.06.020. Epub 2015 Jul 17. PMID 26194770
- [Background] Jasin ME. Nonsurgical rhinoplasty using dermal fillers. Facial Plast Surg Clin North Am. 2013 May;21(2):241-52. doi: 10.1016/j.fsc.2013.02.004. PMID 23731585
- [Background] Nguyen PS, Baptista C, Casanova D, Bardot J, Magalon G. [Autologous fat grafting and rhinoplasty]. Ann Chir Plast Esthet. 2014 Dec;59(6):548-54. doi: 10.1016/j.anplas.2014.05.006. Epub 2014 Jul 3. French. PMID 24997796
- [Background] Adamson PA, Warner J, Becker D, Romo TJ 3rd, Toriumi DM. Revision rhinoplasty: panel discussion, controversies, and techniques. Facial Plast Surg Clin North Am. 2014 Feb;22(1):57-96. doi: 10.1016/j.fsc.2013.09.002. PMID 24290995
- [Background] Xu J, Jiang B, Shen Y. Effectiveness of Autologous Fat Grafting in Scaring After Augmentation Rhinoplasty. J Craniofac Surg. 2019 May/Jun;30(3):914-917. doi: 10.1097/SCS.0000000000005248. PMID 31048617
- [Background] Cakir B, Oreroglu AR, Daniel RK. Surface Aesthetics in Tip Rhinoplasty: A Step-by-Step Guide. Aesthet Surg J. 2014 Aug;34(6):941-55. doi: 10.1177/1090820X14537643. Epub 2014 Aug 1. PMID 24936094